CLINICAL TRIAL: NCT07071766
Title: Adaptation and Implementation of an Evidence-Based Parenting Intervention for Postpartum Women Receiving Medications for Opioid Use Disorder
Brief Title: Improving Outcomes for Early Postpartum Mothers in Outpatient MOUD Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 287138
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-04

CONDITIONS: Substance Use Treatment; Perinatal Substance Use; Parenting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Baby & Me (Experimental): Baby & Me is a manualized parenting education program originally developed for the use in the Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) offices in Arkansas. The program is designed to promote child well-being, reduce parental stress, and prevent child abuse and neglect among WIC recipients who are in their third trimester of pregnancy or have a newborn up to one-month of age. The program is delivered individually to new parents and caregivers via monthly 30-minute sessions over seven months and aims to ensure that new parents and caregivers receive evidence-based parenting education relevant to safe sleep practices, responding to infant cries, maternal mood and self-care, home safety, and developmental milestones. The original Baby & Me curricula was adapted to be delivered in outpatient substance use treatment settings to newly postpartum women receiving medications for opioid use disorder (MOUD) for this study.
  Interventions: Behavioral: Proud of Baby and Me

INTERVENTIONS:
Behavioral: Proud of Baby and Me — The original Baby & Me curricula was adapted to be delivered in outpatient substance use treatment settings to newly postpartum women receiving medications for opioid use disorder (MOUD) for this study.

SUMMARY:
Drug overdose is a leading cause of death among postpartum women and opioid-related mortality is 4 times higher in the postpartum period when compared to the third trimester of pregnancy. Medications for opioid use disorder (MOUD; e.g., methadone or buprenorphine) are the recommended standard of care for perinatal women with OUD. Studies indicate that 50-60% of perinatal women with OUD initiate medications during pregnancy; however, over half will prematurely discontinue treatment within the first six months of childbirth due to stressors experienced in the postpartum period. Common stressors that contribute to MOUD treatment discontinuation in this population are return to opioid use, mental health symptoms including depression, parenting-related stressors such as challenges in infant care and bonding, Neonatal Abstinence Syndrome (NAS), child welfare involvement, and feelings of guilt, shame, and stigma. Thus, there is an urgent need to develop effective, recovery-oriented support interventions that promote the initiation and continuity of MOUD treatment in the postpartum period. The current study utilizes community-engaged research methods to identify and prioritize the early parenting-related needs of postpartum women receiving MOUD to inform the adaptation and implementation of an evidence-based parenting intervention for this population receiving outpatient treatment for opioid use disorder.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Understand and speak English
* Able to give informed consent
* Receiving medications for opioid use disorder in the outpatient clinical setting
* Between 28 weeks gestation and up to 12 months postpartum

Exclusion Criteria:

* Unwilling to consent
* Before 28 weeks gestation and beyond 12 months postpartum at enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 10 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Program Utilization | Up to 12 months after delivery
  % of eligible women who choose to enroll in Baby & Me
Program Acceptability | Up to 12 months after delivery
  Self-report ratings of the acceptability of Proud of Baby & Me
Client Satisfaction | Up to 12 months after delivery
  Self-reported scores on the Client Satisfaction Questionnaire

SECONDARY OUTCOMES:
Depressive Symptoms | Up to 12 months after delivery
  Self-report scores of the Edinburg Postnatal Depression Scale
Parental Stress | Up to 12 months after delivery
  Self-reported scores on the Parenting Stress Index - Short Form
Parenting Confidence | Up to 12 months after delivery
  Self-reported scores of perceived parenting confidence on the Karitane Parenting Confidence Scale

OTHER OUTCOMES:
Drug Use and Cravings | Up to 12 months after delivery
  Self-reported drug use and cravings using the NIDA Modified ASSIST

CONTACTS AND LOCATIONS:
Overall Officials: Mollee K Steely Smith, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No